CLINICAL TRIAL: NCT03492853
Title: The Association of the Peripheral Retinal Changes and Genotypic Changes in Patients With Age Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Tamara Knezevic, medical doctor, ophthalmologist, University Hospital Sestre Milosrdnice
Other Study IDs: UHSestre1
Record Dates: First submitted 2018-04-02; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Peripheral Retinal Degenerations, Age Related Macular Degeneration Polymorphisms
MeSH Terms: interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The DNA was extracted from peripheral blood and then sequenced for SNP's.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with AMD: 150 patients with age related macular degeneration more than 50 years old who will have retina photodocumented and genotyped for AMD SNP's
  Interventions: Genetic: DNA extraction and sequencing
- control group: 150 patients in control group without the clinical signs of the disease more than 50 years old who will have retina photodocumented and genotyped for AMD SNP's
  Interventions: Genetic: DNA extraction and sequencing

INTERVENTIONS:
Genetic: DNA extraction and sequencing — DNA extraction from peripheral blood and KASP sequencing

SUMMARY:
Purpose: To examine the genotypes associated with the peripheral retinal phenotypic features in patients with age-related macular degeneration documented with wide-field imaging.

Design: Clinic-based case series study in Croatia. Participants: 160 patients >50 years of age known to have early or advanced AMD and 150 subjects >50 years of age without known AMD (controls) Methods: Both groups of patients were examined with ophthalmoscopy and OCT to confirm their classification. Posterior and peripheral fundus features were documented with Optos wide-field imaging (Optos P200MA, Optos Plc, Dunfermline, Scotland) and graded. DNA was extracted from blood samples and gene polymorphisms were evaluated for complement factor H (CFH) rs1061170 and rs1410996, age-related maculopathy susceptibility (ARMS2) rs10490924, high temperature requirement factor A1 (HtrA1) rs11200638, complement factor B (CFB) rs4151667 and rs641153, complement factor 2 (C2) rs9332739 and rs547154 and complement factor 3 (C3) rs2230199.

DETAILED DESCRIPTION:
Purpose: To examine the genotypes associated with the peripheral retinal phenotypic features in patients with age-related macular degeneration documented with wide-field imaging.

Design: Clinic-based case series study in Croatia. Participants: Using standard protocols, 160 patients >50 years of age known to have early or advanced AMD and 150 subjects >50 years of age without known AMD (controls) were studied.

Materials and methods: Both groups of patients were examined with ophthalmoscopy and OCT to confirm their classification. Posterior and peripheral fundus features were documented with Optos wide-field imaging (Optos P200MA, Optos Plc, Dunfermline, Scotland) and graded. DNA was extracted from blood samples and gene polymorphisms were evaluated for complement factor H (CFH) rs1061170 and rs1410996, age-related maculopathy susceptibility (ARMS2) rs10490924, high temperature requirement factor A1 (HtrA1) rs11200638, complement factor B (CFB) rs4151667 and rs641153, complement factor 2 (C2) rs9332739 and rs547154 and complement factor 3 (C3) rs2230199.

The study cohort was identified among the clinical patients at the University Department of Ophthalmology at University Hospital Centre "Sestre milosrdnice", Zagreb, Croatia. The protocol was approved by the Ethics Committee approval (EP-13030/11-13) of the University Hospital Centre "Sestre milosrdnice" and complied with the tenets of the Declaration of Helsinki with the informed consent obtained from all the participants. We included 160 subjects in AMD group and 150 subjects in the control group who met the following criteria: age exceeding 50 years, clinical signs of AMD in at least one eye in AMD group and without signs of the disease in the control group. Exclusion criteria were as follows: confounding maculopathy of any etiology, having a myopic refractive error more than -3.0 diopters in either eye, failure to obtain readable color images documenting at least 270 degrees of the retina (three quadrants), or failure to provide a peripheral blood sample for DNA extraction. All the participants were examined according to standardized examination protocols where the macular region and retinal periphery were photodocumented with Resmax and wide field imaging respectively using the Optos P200MA camera (Optos plc, Dumfermline Scotland).23 Phenotypes Eligibility for the AMD group was determined according to an international classification of AMD.24,25 The retinal periphery was defined as an extramacular area 6000 µm diameter distant from the foveolar centre and a grid template was used for measuring the distance. Following peripheral retinal phenotypes were documented: peripheral drusen, reticular pigmentations (RP), hyperpigmentations (pigment clumping (PC) or nevus (N)), hypopigmentations (peripheral retinal pigment defects (RPD) or atrophic areas (AA)), other degenerations in aggregate (OD) which include any of the following: microcystoid degenerations with degenerative retinoschisis (RD), lattice degenerations (LD), snail-track degeneration (ST), white-without pressure (WWP), paving stone degeneration(also known as cobblestone) (PS), retinal holes (R) and vitreal opacities (VO). The inclusion criteria for the peripheral retinal change was its size which had to exceed at least one hour of the retinal periphery Main outcome measures: The type, localization and frequency of peripheral retinal changes and gene polymorphisms of participants in both groups were examined.

ELIGIBILITY:
Inclusion Criteria:

* in AMD group-patients with the signs of AMD disease

Exclusion Criteria:

* confounding maculopathy of any etiology, having a myopic refractive error more than -3.0 diopters in either eye, failure to obtain readable color images documenting at least 270 degrees of the retina (three quadrants), or failure to provide a peripheral blood sample for DNA extraction

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included 160 subjects in AMD group and 150 subjects in the control group who met the following criteria: age exceeding 50 years, clinical signs of AMD in at least one eye in AMD group and without signs of the disease in the control group. Exclusion criteria were as follows: confounding maculopathy of any etiology, having a myopic refractive error more than -3.0 diopters in either eye, failure to obtain readable color images documenting at least 270 degrees of the retina (three quadrants), or failure to provide a peripheral blood sample for DNA extraction. All the participants were examined according to standardized examination protocols where the macular region and retinal periphery were photodocumented with Resmax and wide field imaging respectively using the Optos P200MA camera (Optos plc, Dumfermline Scotland).
Sampling Method: Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
the association of the peripheral retina changes and genotyping | 2 years
  the association between those two parameters

IPD SHARING:
Plan to Share IPD: No